CLINICAL TRIAL: NCT03330561
Title: A Phase 1, Open-Label, Dose Escalation Study of PRS-343 in Patients With HER2-Positive Advanced or Metastatic Solid Tumors
Brief Title: PRS-343 in HER2-Positive Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pieris Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRS-343-PCS_04_16
Record Dates: First submitted 2017-10-19; First posted 2017-11-06 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: HER2-positive Breast Cancer; HER2-positive Gastric Cancer; HER2-positive Bladder Cancer; HER2-positive Solid Tumor
Keywords: HER2-positive breast cancer; HER2 -positive gastric cancer; HER2-positive bladder cancer; Pieris; PRS-343; Anticalin; Bi-specific; 4-1BB; CD137; HER2

STUDY DESIGN:
Intervention Model Description: Drug PRS-343 Monotherapy
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRS-343 (Experimental)
  Interventions: Drug: PRS-343

INTERVENTIONS:
Drug: PRS-343 — PRS-343
  Other Names: HER2/41BB Bispecific

SUMMARY:
A multi center, open-label, Phase 1 dose escalation study with expansion cohort is designed to determine the MTD, RP2D and dosing schedule of PRS-343 in patients with HER2+ advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
The study will evaluate PRS-343 administered by intravenous (IV) infusion every 3 weeks (Schedule 1) initially. If safety, PK, and PD data suggest a different dosing schedule should be evaluated, Schedule 2 and/or 3 (dosing every 2 weeks in a 28-day cycle or once a week in a 21-day cycle, respectively) may be conducted. Separate MTDs may be determined for each schedule evaluated. Dose-limiting toxicities (DLTs) will be reported during the first cycle of each schedule (e.g., 21 days after the first dose in Cycle 1 for Schedule 1). Patients will be monitored for safety throughout the study. Dosing will continue until criteria for study drug discontinuation are met (disease progression or withdrawal from the study).

Patients with unknown HER2 status will be consented separately in a pre-screening visit in order to undergo HER2 testing prior to screening. All patients will be evaluated at screening (Day 28 to 1) and baseline (Day 1 predose).

Once the MTD has been established, up to 30 additional patients with locally advanced or metastatic HER2+ solid tumors considered likely to respond to a HER2 targeted CD137 agonist (e.g. gastric/gastroesophageal/esophageal, breast, bladder) may be enrolled in individual expansion cohorts. The expansion cohort will be enrolled at the MTD and/or at a lower dose level if safety/PD/PK/efficacy data support further evaluation of a lower dose level in order to determine the RP2D. The RP2D may be equivalent to or lower than the MTD.

An End-of-Treatment Visit will be performed at the time of treatment discontinuation. Patients will be evaluated 30 days after the End-of-Treatment Visit or prior to starting subsequent therapy, if sooner, at the Safety Follow-up Visit to assess any ongoing AEs as outlined in the protocol.

Obinutuzumab pre-treatment cohorts: The potential of obinutuzumab pre-treatment to reduce formation of ADA will be studied in a cohort of up to ten patients receiving PRS-343 at a dose of 8 mg/kg Q2 weeks (corresponding to Cohort 11b).

Patients will be assessed for tumor response/progression per RECIST v1.1

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent obtained prior to performing any study procedure, including pre-screening and screening procedures.
2. Men and women ≥18 years.
3. Dose escalation: Histologically or cytologically confirmed diagnosis of unresectable/locally advanced and/or metastatic HER2+ solid tumor malignancy and for which standard therapies are not available, are no longer effective, are not tolerated, or have been declined by the patient.

   Expansion cohort: Locally advanced or metastatic HER2+ solid tumors considered likely to respond to a HER2-targeted CD137 agonist (e.g. gastric/gastroesophageal/esophageal, breast, bladder).
4. Dose escalation and expansion cohort: HER2+ tumors documented by clinical pathology report:

   1. Assessment of HER2 status in patients with breast cancer should follow the 2013 American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) criteria (37) as practicable.
   2. Assessment of HER2 status in patients with gastric and gastroesophageal junction adenocarcinoma should follow the criteria published by Ruschoff et al. (38) as practicable.
   3. Assessment of HER2 status in patients with non-breast/non-gastric cancers may follow local institutional criteria. These criteria should be made available to the Sponsor.
   4. All patients with breast and gastric/gastroesophageal junction cancers should have HER2 testing performed using a FDA approved test in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory.
   5. Patients for whom the clinical pathology report includes only IHC as 3+ (does not reflex to ISH) may enroll without written report of ISH determined HER2 copy number, provided the investigational site confirms that archival tissue is available.
5. Patients with breast cancer and gastric and gastroesophageal junction cancer must have received at least 1 prior HER2 targeted therapy for advanced/metastatic disease.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
7. Estimated life expectancy of at least 3 months.
8. Measurable disease according to RECIST v1.1.
9. Adequate organ function as defined below:

   1. Serum AST and ALT ≤ 3 X ULN
   2. Total serum bilirubin ≤ 1.5 X ULN
   3. Serum creatinine ≤ 1.5 X ULN OR calculated glomerular filtration rate (GFR) by Cockcroft-Gault formula ≥ 50 mL/min
   4. Hemoglobin ≥ 9 g/dL
   5. ANC ≥ 1500/mm3
   6. Platelet count ≥ 75,000/mm3
   7. Left ventricular ejection fraction (LVEF) determined by echocardiogram or multi-gated acquisition scan ≥ 50%
10. Any prior cumulative doxorubicin dose must be ≤ 360 mg/m2; prior cumulative epirubicin dose must be ≤ 720 mg/m2.
11. Women of childbearing potential must have a negative serum or urine pregnancy test within 96 hours prior to start of study drug.
12. Women must not be breastfeeding.
13. Women of childbearing potential must agree to follow instruction for method(s) of contraception for the duration of treatment with study drug PRS-343 plus 90 days post-treatment completion.
14. Males who are sexually active with women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug PRS 343 plus 90 days post-treatment completion.

Exclusion criteria:

1. Known uncontrolled central nervous system (CNS) metastases and/or carcinomatous meningitis. Note: Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are clinically stable off steroids for at least 7 days prior to study treatment. Carcinomatous meningitis precludes a patient from study participation regardless of clinical stability.
2. History of acute coronary syndromes, including myocardial infarction, coronary artery bypass graft, unstable angina, coronary angioplasty or stenting within past 24 weeks.
3. History of or current Class II, III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system (Appendix B).
4. History of ejection fraction drop below the lower limit of normal with trastuzumab and/or pertuzumab.
5. Medical, psychiatric, cognitive or other conditions that compromise the patient's ability to understand the patient information, to give informed consent, to comply with the study protocol or to complete the study.
6. Any severe concurrent disease or condition (includes active infections, cardiac arrhythmia, interstitial lung disease) that in the judgment of the investigator would make study participation inappropriate for the patient.
7. Previously known infection with human immunodeficiency virus (HIV); or hepatitis B or hepatitis C infection. Patients with positive hepatitis B core antibody (HBcAb) require assessment and monitoring of virus deoxyribonucleic acid (DNA) status; patients with positive hepatitis C virus (HCV) core antibody can enroll if HCV ribonucleic acid (RNA) is negative. Patients with latent or active hepatitis B infection are excluded from the pre-treatment Cohort receiving obinutuzumab.
8. History of infusion reactions to any component/excipient of PRS-343.
9. Systemic steroid therapy (>10 mg daily prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment (Note: topical, inhaled, nasal and ophthalmic steroids are not prohibited). This criterion does not apply to patients receiving obinutuzumab as pre-treatment.
10. Autoimmune disease that has required systemic treatment in the past (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed.
11. Has not recovered from the adverse effect of previous anticancer treatments to pre-treatment baseline or Grade 1 except for alopecia, anemia (hemoglobin must meet the study inclusion criteria) and peripheral neuropathy (which must have recovered to ≤ Grade 2) nausea and diarrhea if anti-emetic and anti-diarrheal treatment has not been exhausted.
12. History of a second primary cancer with the exception of 1) curatively treated non-melanomatous skin cancer, 2) curatively treated cervical or breast carcinoma in situ, or 3) other malignancy with no known active disease present and no treatment administered during the last 2 years.
13. Receipt of investigational treatment within 3 weeks of scheduled Cycle 1 Day 1 (C1D1) dosing.
14. Receipt of cytotoxic chemotherapy within 3 weeks (6 weeks for nitrosoureas and mitomycin C) of scheduled C1D1 dosing.
15. Receipt of radiation therapy within 3 weeks of scheduled C1D1 dosing, unless the radiation comprised a limited field to non-visceral structures (e.g., limb bone metastasis).
16. Receipt of treatment with immunotherapy, biological therapies, targeted small molecules, hormonal therapies within 3 weeks of scheduled C1D1 dosing.
17. Receipt of trastuzumab or ado-trastuzumab emtansine or any other experimental drug that engages the same epitope as trastuzumab within 4 weeks of scheduled C1D1 dosing.
18. Concurrent enrollment in another therapeutic clinical trial.
19. Major surgery within 3 weeks of scheduled C1D1 dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of AEs graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03 | Up to 36 months

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Up to 36 months
Area under the plasma concentration versus time curve (AUC) | Up to 36 months
Time to maximum dose concentration (Tmax) | Up to 36 months
Terminal half life (t1/2) | Up to 36 months
Tumor responses as defined by the Response Evaluation in Solid Tumors (RECIST) v.1.1 | Up to 36 months
Duration of response | Up to 36 months
Disease control rate | Up to 36 months
Presence of PRS-343 anti-drug antibodies | Up to 36 months
Biomarkers (CD137, soluable HER2, cell surface antigens for immunotyping) in tumor tissues and blood samples | Up to 36 months

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of California Los Angeles (UCLA), Santa Monica, California
  - Georgetown University, Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - M.D. Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - START - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided